CLINICAL TRIAL: NCT03475407
Title: The Effects of Intravitral Ozurdex Implant in DME: Cytokine Change in Aqueous Humor
Brief Title: The Effects of Intravitreal Ozurdex Implant in DME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nune Eye Hospital, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Oh Woong Kwon, Chief of retina center in Nune Eye Hospital, Nune Eye Hospital, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRBF004
Record Dates: First submitted 2015-04-14; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; cytokine; dexamethasone
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Group (Experimental): Ozurdex intravitreal injection
  Interventions: Drug: Ozurdex intravitreal injection

INTERVENTIONS:
Drug: Ozurdex intravitreal injection — 1. Ozurdex intravitreal injection and Antreior Chamber(AC) paracentesis at baseline
  2. AC paracentesis at 6 wk
  3. intravitreal Ozurdex injection and AC paracentesis at 18wk or 24wk

SUMMARY:
Intravitreal Ozurdex implant therapy improves visual outcome and OCT findings. The purpose of this study is that these results are correlated with the change of cytokine level known to be increased in DME patients.

ELIGIBILITY:
Inclusion Criteria:

The patients of Type 1 or Type 2 Diabetes Mellitus fulfilling the following inclusion criteria shall be enrolled in the study:

* Patients of Non Proliferative Diabetic Retinopathy(NPDR) with clinically significant macular edema(CSME)
* Patients with Proliferative Diabetic Retinopathy(PDR) with CSME where proliferative component has been adequately treated with laser photocoagulation
* Diabetic patients with cystoids macular edema
* Minimum central thickness on OCT not less than 300 microns
* BCVA 20/30~20/320

Exclusion Criteria:

* Patients with history of Anti-VEGF or steroid injection, any type of laser treatments, vitrectomy, cataract surgery within 6 months
* Patients with history of ocular hypertension or glaucoma
* Patients with media haze or pupillary non-dilation that does not allow good fundus photography, FFA and OCT
* Patients with macular ischemia on FFA
* Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva
* Patients whose posterior lens capsule is not intact.
* patients with known hypersensitivity to any components of this product.
* patients with vitreous hemorrhage
* patients who have systemic treatment effect on study results
* patients who enrolled other clinical study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Central foveal thickness(CFT, height in micrometers) | Baseline, 1 week, 6 weeks, 12 weeks, 18 weeks, 24 weeks

SECONDARY OUTCOMES:
Changes of aqueous humor cytokine (VFGF, IL-2, IL-6,IL-8, MCP-1) | Baseline, 6 weeks, 18 weeks
Changes of Best corrected Visual acuity(BCVA, ETDRS scale) | Baseline, 1 week, 6 weeks, 12 weeks, 18 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oh Woong Kwon, MD PhD, Principal Investigator — Nune Eye Hospital
Locations (1):
- Nune Eye Hospital, Seoul, South Korea